CLINICAL TRIAL: NCT05355870
Title: mHealth Cognitive Training Intervention Pilot for Older Chinese Americans
Brief Title: Cognitive Training RCT for Older Chinese Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: New York University (Other); National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00109934; R21AG075228 (NIH)
Record Dates: First submitted 2022-04-21; First posted 2022-05-02 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-01

CONDITIONS: Cognitive Health; mHealth Application; Experience-based Co-design; Cognitive Training; Ethnogeriatrics
Keywords: mHealth; Cognitive Training; Pilot; Chinese Americans

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Training (Experimental): Participants in the experimental arm will be provided a brochure that included information on basic knowledge of ADRD, signs and symptoms related to ADRD, the definition and the potential benefits of cognitively stimulating activities in maintaining cognitive function, and examples of cognitively stimulating activities.
  Participants in this arm will complete a series of cognitive training exercises on a smartphone/tablet. The anticipated training will last for 12 weeks and involve 3-4 sessions per week (20-30 min/ session).
  Interventions: Behavioral: Cognitive Training Intervention
- Passive Control (No Intervention): A passive control group will be included in this pilot trial. Participants in this passive control arm will be provided a brochure that included information on basic knowledge of ADRD, signs and symptoms related to ADRD, the definition and the potential benefits of cognitively stimulating activities in maintaining cognitive function, and examples of cognitively stimulating activities.

INTERVENTIONS:
Behavioral: Cognitive Training Intervention — Participants in the intervention group will complete a series of cognitive training exercises adapted from the BrainHQ. Results from the intervention development activities will be used to finalize the dose, frequency, and duration of the training. Each session will include 2 training exercises that target different cognitive domains. As participants progress, the difficulty level will be automatically adapted based on participants' performance.
  Arms: Cognitive Training

SUMMARY:
The purpose of this study is to develop and pilot test a mHealth intervention for cognitive training that is culturally and linguistically relevant to older Chinese Americans

DETAILED DESCRIPTION:
This is an NIH Stage 1 pilot randomized controlled trial. The purpose of this trial is to evaluate the feasibility, acceptability, and obtain preliminary effect sizes on outcomes of a cognitive training intervention. The cognitive training intervention will be app-based and will be co-developed with older Chinese Americans and adult children to ensure it is culturally and linguistically relevant.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Chinese
* are age 60 or older
* are fluent in written and spoken Chinese and/or English
* have the visual capacity to read a smartphone or a tablet screen and have the auditory capacity to understand normal speech
* have no self-reported diagnosis of ADRD or cognitive impairment, and are capable of making an informed consent

Exclusion Criteria:

* Individuals are excluded if they are bed-ridden
* receiving chemotherapy for malignancy
* have other life-threatening illnesses

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Feasibility as Measured by the status of study accrual | Approximately 6 months
  Meeting the recruitment goal of 30 eligible participants in 6 months (Yes/No)
Feasibility as Measured by Study Adherence | 12 weeks
  The proportion of participants in the intervention arm who successfully completing all intervention sessions
Feasibility as Measured by Adherence to Measurement Strategies at week 8 | 8 weeks
  The proportion of participants completing the 8-week assessments in both arms
Feasibility as Measured by Adherence to Measurement Strategies at week 12 | 12 weeks
  The proportion of participants completing the 12-week assessments in both arms
Acceptability as Measured by the Client Satisfaction Questionnaire | 12 weeks
  The Client Satisfaction Questionnaire (CSQ) ranges from 8 to 32, with scores over the 80% suggested adequate acceptability
Duration of cognitive training as Measured by the average time to complete a cognitive exercise | Over the course of the intervention, 12 weeks
  The average time in minutes to complete a cognitive exercise for participants in the intervention arm over the course of study participation, with longer duration indicated longer training
Days of App use as Measured by the percentage of days that participants use the app | Over the course of the intervention, 12 weeks
  The percentage of days that participants use the app for participants in the intervention arm over the course of study participation, with higher proportion indicated more days engaged in cognitive training
Change in Global cognition as a composite measure of Mini-Mental State Examination(MMSE), Digit Span Test, verbal fluency, and the Trail Making Test | Baseline, 8 weeks, 12 weeks
  A z-score of each test will be calculated and the average z-score that ranges from -1 to 1 will be used to measure global cognition, with higher score indicated better cognitive function

SECONDARY OUTCOMES:
Change in Loneliness as Measured by the University of California, Los Angeles three item Loneliness Scale | Baseline, 8 weeks, 12 weeks
  The University of California, Los Angeles (UCLA) Loneliness Scale ranges from 3 to 9, with higher scores indicated greater degrees of loneliness
Change in Anxiety as Measured by the Hospital Anxiety and Depression Scale-Anxiety Subscale | Baseline, 8 weeks, 12 weeks
  The HADS - Anxiety Scale ranges from 0 to 21, with higher scores indicated greater degrees of anxiety
Change in Depressive Symptoms as Measured by the Patient Health Questionnaire-9 | Baseline, 8 weeks, 12 weeks
  PHQ-9 ranges from 0 to 27, with higher scores indicated greater depressive symptoms
Change in Quality of Life as Measured by the World Health Organization Quality of Life Instrument- Abbreviated Version (WHOQOL-BREF) | Baseline, 8 weeks, 12 weeks
  The WHOQOL-BREF ranges from 0 to 100, with higher scores indicated better quality of life
Change in Physical Functioning as Measured by the Activities of Daily Living and Instrumental Activities of Daily Living Scale | Baseline, 8 weeks, 12 weeks
  Score ranges from 14 to 52, with higher scores indicated higher degree of physical functioning

CONTACTS AND LOCATIONS:
Overall Officials: Hanzhang Xu, PhD, Principal Investigator — Duke University
Locations (1):
- North Carolina (Participants Homes), Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xue T, Wei AA, Wu B, Sanders C, McConnell ES, Xu H. Co-Designed Mobile-Based Cognitive Training for Older Chinese Americans: Protocol for a Pilot Randomized Controlled Trial Assessing Feasibility and Acceptability. JMIR Res Protoc. 2025 Jul 21;14:e69303. doi: 10.2196/69303. PMID 40690756

DOCUMENTS (1):
  • Informed Consent Form (2025-01-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT05355870/ICF_000.pdf